CLINICAL TRIAL: NCT04498585
Title: Virtual Reality Stimulation to Relax and Reduce the Incidence of Delirium
Brief Title: Virtual Reality to Reduce Delirium
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Decreased resources due to COVID-19
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: KEK2020-00039; 2020-00039 (Other: Ethics Committee of the Canton of Bern)
Record Dates: First submitted 2020-07-28; First posted 2020-08-04 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Delirium; Cognitive Impairment
Keywords: Virtual Reality; Delirium; Intensive Care Unit; Critical Care; Movement Analysis
MeSH Terms: conditions — Delirium; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants who will be receiving standard ICU care and additionally the VR stimulation during their ICU stay.
  Interventions: Other: VR Stimulation
- Control (No Intervention): Patients in the ICU who will be receiving standard ICU care during their ICU stay. Participants in this arm will not be receiving VR stimulation.

INTERVENTIONS:
Other: VR Stimulation — Participants in the intervention group will be provided with 30 minutes of relaxing, 360-degree virtual reality stimulation and corresponding sounds, three times a day (morning, midday, evening) everyday during their stay in the ICU, up to a maximum of 14 days.
  Other Names: Visuo-acoustic stimulation
  Arms: Intervention

SUMMARY:
Delirium has been long considered as a major contributor to cognitive impairments following a critical illness. Currently, both pharmacologic and non-pharmacologic prevention and treatment strategies are used in the intensive care unit, despite these strategies remaining controversial. However, with previous studies showing the feasibility of using virtual reality (VR) within the critical care setting, the investigators propose to use this technology to investigate the effect of 360-degree immersive virtual reality stimulation on the incidence of delirium in the ICU.

Stimulation will be provided for 30 minutes, three times a day, evenly spaced between 7:00 AM and 7:00 PM, using a commercially available head-mounted display. The investigators hypothesize that by providing relaxing virtual environments to patients through a head-mounted display and headphones, the incidence of delirium will be lower compared to the control group receiving no VR stimulation. Secondary outcomes will include evaluating the movement patterns and intensity between the intervention and control group, and between patients with and without delirium, using inertial measurement units and an under mattress bed sensor. It is hypothesized that it will be possible to detect difference in movement patterns between groups and identify patterns indicating the presence or absence of delirium. Secondary objective also include the evaluation of the effect of VR on duration of delirium. Here it is hypothesized that the duration of delirium will be shorter in participants receiving the VR stimulation compared to those in the control group. Physiological parameters (e.g. heart rate, respiration rate, oxygen saturation, etc.) will also be recorded during the stimulation to further understand what, if any, effect VR has.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent (by the patient, relatives, or authorized representative)
* No severe visual or auditory impairments (strabismus, macular degeneration, retinopathy)
* Estimated length of stay >24 hours
* Can keep eyes open for at least 30 seconds
* German or French speaking

Exclusion Criteria:

* Known psychotic disorders associated with delusions (e.g. schizophrenia)
* Recent history of major depression
* Admission for drug overdose

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self identified gender
Enrollment: 920 (Estimated)
Dates: Start 2021-04-14 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Delirium | Number of incidences during stay in the intensive care unit (to a maximum of 14 days)
  Delirium will be assessed 3 times a day using the Intensive Care Delirium Screening Checklist. The screening will be conducted by trained critical care nurses. If a score greater than or equal to 4 is recorded, this will count as an incidence of delirium.

SECONDARY OUTCOMES:
Pattern of the movements before and during delirium | Recorded during entire stay in the ICU (to a maximum of 14 days)
  Movement patterns, measured as acceleration and rotation, will be measured using inertial measurement units. The data will be used to determine if there is a change in pattern or intensity between periods before and during delirium.
Intensity of the movements before and during delirium | Recorded during entire stay in the ICU (to a maximum of 14 days)
  Movement patterns, measured as acceleration and rotation, will be measured using inertial measurement units. The data will be used to determine if there is a change in intensity between periods before and during delirium.
Duration of Delirium | Recorded during entire stay in the ICU (to a maximum of 14 days)
  The duration of delirium will be evaluated per 8 hour periods, or as needed, while patients are in the ICU. If the participant is assessed as delirious during any of the assessments during an 8 hour span, the entire period will count as delirious.

OTHER OUTCOMES:
Cognitive Functioning | Compared between functioning at discharge to 6-months post-discharge.
  Cognitive abilities will be measured using the Montreal Cognitive Assessment (MoCA).
Health Related Quality of Life | Compared between quality pre-admission to 6-months post-discharge.
  Quality of life is examined via the EQ-5D questionnaire (official name, not abbreviated). The five-level version (5L) will be used. The five levels of the scale, scored from 1 to 5 are: no problems, slight problems, moderate problems, severe problems, unable to/extreme problems. The numbers for the five dimensions are subsequently combined to create a unique 5-digit code which represents the respondent's overall health state. This means an index of 11111 is the best possible health, and 55555 is the worst possible health.
Functional Independence | Compared between quality pre-admission to 6-months post-discharge.
  Independence is examined using the Functional Independence Measure (FIM).
Heart Rate | Every stimulation period for the duration of the patient's time in the ICU (to a maximum of 14 days).
  Changes in heart rate (beats per minute) recorded from the patient will be compared from the start of the stimulation to the end of the stimulation period.
Blood Pressure | Every stimulation period for the duration of the patient's time in the ICU (to a maximum of 14 days).
  Changes in blood pressure (mmHg) recorded from the patient will be compared from the start of the stimulation to the end of the stimulation period.
Respiration Rate | Every stimulation period for the duration of the patient's time in the ICU (to a maximum of 14 days).
  Changes in respiration rate (breaths per minute) recorded from the patient will be compared from the start of the stimulation to the end of the stimulation period.
Oxygen Saturation | Every stimulation period for the duration of the patient's time in the ICU (to a maximum of 14 days).
  Changes in oxygen saturation (%) recorded from the patient will be compared from the start of the stimulation to the end of the stimulation period.
System Usability Scale | Once a day for the duration of the patient's time in the ICU (to a maximum of 14 days).
  The 10-item System Usability Scale is used to collect data on the user's (nurse providing VR stimulation) subjective usability assessments. There are five response options per question; from Strongly disagree (1) to Strongly agree (5). For each odd numbered question, subtract 1 from the score. For each even numbered question, subtract the score from 5. Add up the new values calculated and multiply this total by 2.5. This gives a final score from 0 - 100 (this is not a percentage, but values can be normalized to produce a percentile ranking). A score above 68 is considered above average, and below 68 is below average.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Hänggi, Dr. med, Principal Investigator — Department of Intensive Care Medicine, University Hospital Bern (Inelspital)
Locations (1):
- Inselspital, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The investigators will ask patients to provide informed consent for sharing their anonymized data. Once the study results are published, the investigators will make the de-identified study dataset available for secondary analyses by sharing the dataset upon reasonable request.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data will be shared once study results have been published.
Access Criteria: To be determined.

REFERENCES:
- [Background] Chanques G, Ely EW, Garnier O, Perrigault F, Eloi A, Carr J, Rowan CM, Prades A, de Jong A, Moritz-Gasser S, Molinari N, Jaber S. The 2014 updated version of the Confusion Assessment Method for the Intensive Care Unit compared to the 5th version of the Diagnostic and Statistical Manual of Mental Disorders and other current methods used by intensivists. Ann Intensive Care. 2018 Mar 1;8(1):33. doi: 10.1186/s13613-018-0377-7. PMID 29492696
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Santos E, Cardoso D, Neves H, Cunha M, Rodrigues M, Apostolo J. Effectiveness of haloperidol prophylaxis in critically ill patients with a high risk of delirium: a systematic review. JBI Database System Rev Implement Rep. 2017 May;15(5):1440-1472. doi: 10.11124/JBISRIR-2017-003391. PMID 28498176
- [Background] Pandharipande PP, Girard TD, Ely EW. Long-term cognitive impairment after critical illness. N Engl J Med. 2014 Jan 9;370(2):185-6. doi: 10.1056/NEJMc1313886. No abstract available. PMID 24401069
- [Background] Girard TD, Exline MC, Carson SS, Hough CL, Rock P, Gong MN, Douglas IS, Malhotra A, Owens RL, Feinstein DJ, Khan B, Pisani MA, Hyzy RC, Schmidt GA, Schweickert WD, Hite RD, Bowton DL, Masica AL, Thompson JL, Chandrasekhar R, Pun BT, Strength C, Boehm LM, Jackson JC, Pandharipande PP, Brummel NE, Hughes CG, Patel MB, Stollings JL, Bernard GR, Dittus RS, Ely EW; MIND-USA Investigators. Haloperidol and Ziprasidone for Treatment of Delirium in Critical Illness. N Engl J Med. 2018 Dec 27;379(26):2506-2516. doi: 10.1056/NEJMoa1808217. Epub 2018 Oct 22. PMID 30346242
- [Background] Serafim RB, Bozza FA, Soares M, do Brasil PE, Tura BR, Ely EW, Salluh JI. Pharmacologic prevention and treatment of delirium in intensive care patients: A systematic review. J Crit Care. 2015 Aug;30(4):799-807. doi: 10.1016/j.jcrc.2015.04.005. Epub 2015 Apr 17. PMID 25957498
- [Background] Zayed Y, Barbarawi M, Kheiri B, Banifadel M, Haykal T, Chahine A, Rashdan L, Aburahma A, Bachuwa G, Seedahmed E. Haloperidol for the management of delirium in adult intensive care unit patients: A systematic review and meta-analysis of randomized controlled trials. J Crit Care. 2019 Apr;50:280-286. doi: 10.1016/j.jcrc.2019.01.009. Epub 2019 Jan 12. PMID 30665181
- [Background] Gerber SM, Jeitziner MM, Knobel SEJ, Mosimann UP, Muri RM, Jakob SM, Nef T. Perception and Performance on a Virtual Reality Cognitive Stimulation for Use in the Intensive Care Unit: A Non-randomized Trial in Critically Ill Patients. Front Med (Lausanne). 2019 Dec 10;6:287. doi: 10.3389/fmed.2019.00287. eCollection 2019. PMID 31921867
- [Background] Gerber SM, Jeitziner MM, Wyss P, Chesham A, Urwyler P, Muri RM, Jakob SM, Nef T. Visuo-acoustic stimulation that helps you to relax: A virtual reality setup for patients in the intensive care unit. Sci Rep. 2017 Oct 16;7(1):13228. doi: 10.1038/s41598-017-13153-1. PMID 29038450
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Nasreddine ZS, Phillips NA, Bedirian V, Charbonneau S, Whitehead V, Collin I, Cummings JL, Chertkow H. The Montreal Cognitive Assessment, MoCA: a brief screening tool for mild cognitive impairment. J Am Geriatr Soc. 2005 Apr;53(4):695-9. doi: 10.1111/j.1532-5415.2005.53221.x. PMID 15817019
- [Background] Herdman M, Gudex C, Lloyd A, Janssen M, Kind P, Parkin D, Bonsel G, Badia X. Development and preliminary testing of the new five-level version of EQ-5D (EQ-5D-5L). Qual Life Res. 2011 Dec;20(10):1727-36. doi: 10.1007/s11136-011-9903-x. Epub 2011 Apr 9. PMID 21479777
- [Background] Linacre JM, Heinemann AW, Wright BD, Granger CV, Hamilton BB. The structure and stability of the Functional Independence Measure. Arch Phys Med Rehabil. 1994 Feb;75(2):127-32. PMID 8311667
- [Derived] Naef AC, Jeitziner MM, Gerber SM, Jenni-Moser B, Muri RM, Jakob SM, Nef T, Hanggi M. Virtual reality stimulation to reduce the incidence of delirium in critically ill patients: study protocol for a randomized clinical trial. Trials. 2021 Mar 1;22(1):174. doi: 10.1186/s13063-021-05090-2. PMID 33648572